CLINICAL TRIAL: NCT06992817
Title: Çocuk Judocuların Antrenör Yönlendirmesi ve Eğitim Müdahalelerinin Hidrasyon Durumlarına Etkisi
Brief Title: The Impact of Brief One-time Education and Coach Encouragement on Hydration Status in Child Judo Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Collaborators: Selcuk University (Other); Duzce University (Other); Harran University (Other); Mustafa Kemal University (Other); Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Bayram Ceylan, Assoc. Prof., Kastamonu University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E.912346
Record Dates: First submitted 2025-05-06; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Dehydration in Children; Dehydration
Keywords: hypohydration; health; athletic population; combat sports
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Who Masked: Participant
Masking Description: Athletes were unaware of the intervention conditions assigned to each day, and the educational session was presented without emphasizing its experimental nature. The order of conditions was fixed (control first, then coach encouragement, and finally education) to minimize potential carryover effects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No-intervention (Control) (No Intervention): This arm did not receive any intervention. They completed the training session without any encouragement related to fluid intake.
- Coach encouragement (Intervention 1) (Experimental): During this intervention, athletes were encouraged by their coaches to consume fluids during the training.
  Interventions: Behavioral: Hydration-Coach Encouragement
- Hydration education (Intervention 2) (Experimental): During this interventio, athletes were given a brief hydration education before the training session.
  Interventions: Behavioral: Short Hydration Informative Session

INTERVENTIONS:
Behavioral: Hydration-Coach Encouragement — Athletes were encouraged by their coaches to consume fluids during the training session.
  Other Names: Encouragement
  Arms: Coach encouragement (Intervention 1)
Behavioral: Short Hydration Informative Session — Athletes were given a brief educational session related to importance of hydration before the exercise session.
  Other Names: A brief hydration education
  Arms: Hydration education (Intervention 2)

SUMMARY:
Due to the lack of any comparative study related to effect of different hydration processes, this study aimed to compare the effectiveness of coach encouragement and hydration education in maintaining hydration status in child judo athletes

DETAILED DESCRIPTION:
Forty-seven athletes participated in a four-day training camp, during which hydration status was assessed before and after training sessions under three different conditions: no intervention (control), coach-guided fluid intake encouragement, and pre-training brief one-time hydration education. Athletes were unaware of the intervention conditions assigned to each day, and the educational session was delivered without emphasizing its experimental nature. To minimize potential carryover effects, the sequence of interventions was fixed. Hydration status was objectively monitored using urine specific gravity (USG) and urine color (UC) measurements.

ELIGIBILITY:
Inclusion Criteria:

* having at least three years of judo experience
* having at least a green belt
* being healthy enough to attend all training sessions during the camp.

Exclusion Criteria:

* having less than three years of judo experience
* having orange belt or lower
* not being healthy enough to attend all training sessions during the camp.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
hydration status (i.e., urine specific gravity and urine colour) | 4 days
  A urine sample was taken from each athlete one hour before and immediately after the exercise sessions. The samples were placed in plastic cups and USG was determined with a digital refractometer (ATAGO PAL-10S, Japan) in the training hall by the same researcher each time. USG measurements were carried out after the urine samples were refrigerated to temperature of 20° and UC was classified under LED light condition. As soon as the urine samples were analyzed for USG and classified for urine colour (UC), they were immediately disposed. USG was classified according to suggestion by National Athletic Trainers' Association as hydrated (USG <1.020) and hypohydrated (USG≥1.020).

CONTACTS AND LOCATIONS:
Overall Officials: Şükrü Serdar Balcı, PhD, Principal Investigator — Selcuk University
Locations (1):
- Bartın Judo Hall, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June-September 2025
Access Criteria: Upon request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT06992817/Prot_SAP_000.pdf